CLINICAL TRIAL: NCT00149019
Title: Innovative Approaches for Targeted Immunotherapy of Cancer Using Donor Lymphocytes Labelled With In-vitro Bispecific Antibodies.
Brief Title: Immunotherapy of Cancer Using Donor Lymphocytes Labelled With In-vitro Bispecific Antibodies.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the PI is no longer work at Hadassah
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 240502-HMO-CTIL
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2005-09

CONDITIONS: Metastatic Solid Tumors
MeSH Terms: interventions — Cell- and Tissue-Based Therapy; Antibodies, Bispecific

INTERVENTIONS:
Drug: Cell therapy with bispecific antibodies

SUMMARY:
Patients with resistant metastatic solid tumors failing all conventional modalities who are eligible for immunotherapy by bispecific antibodies.

First step: NST Second step: Patients with tumor cells expressing positive Her-2Neu and/or EpCAM with residual or recurrent disease following NST will be candidates for donor lymphocytes immunotherapy using bispecific antibodies.

Patients with no matched donor available, expressing positive Her-2Neu and/or EpCAM tumor cells, will be eligible for donor mismatched lymphocytes using in-vitro rIL-2 activated allogeneic lymphocytes targeted to the tumor by bispecific antibodies, Her-2Neu and/or EpCAM.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic solid tumors expressing Her-2/Neu or EpCAM, with available match donor for NST.
* Patients with metastatic solid tumors not expected to be cured failing available conventional modalities, age >18, with no upper age limit.
* Patients with metastatic breast cancer failing treatment with Herceptin.
* Patients with metastatic cancer cells expressing Her-2/Neu or EpCAM.
* Patients with evidence of disease following allogeneic stem cell transplantation with tumor cells expressing Her-2/Neu or EpCAM.
* Karnofsky performance status >60%
* Life expectancy > 3 months, to be able to assess response.

Exclusion Criteria:

* Patients not fulfilling any of the above.
* Patients with active or ongoing infection that may endanger their life, whenever immunosuppression may be counter-indicated.
* Pregnant or lactating women.
* Patients positive for HIV.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2002-05; Study Completion 2005-09 (Estimated)

PRIMARY OUTCOMES:
The purpose will be to evaluate safety using donor lymphocytes labelled in-vitro with bispecific antibodies for metastatic cancer patients.

SECONDARY OUTCOMES:
To evaluate primary efficacy using donor lymphocytes labelled in-vitro with bispecific antibodies for metastatic cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel